CLINICAL TRIAL: NCT02822547
Title: Study to Identify Eligible Subjects Using Response Guided Therapy-Stopping Rule for Treatment of Pegylated Interferon Alfa 2a(Pegasys®) in the Korean Chronic Hepatitis B(CHB) Adults.
Brief Title: Study on Treatment of Pegylated Interferon Alfa 2a(Pegasys®) in the Korean Chronic Hepatitis B(CHB) Adults
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Principal Investigator, Sang Hoon Ahn, Professor, Yonsei University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML29378
Record Dates: First submitted 2016-06-30; First posted 2016-07-04 (Estimated); Last update posted 2016-07-04 (Estimated); Status verified 2016-06

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — peginterferon alfa-2a

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Peginterferon alfa-2a (Experimental)
  Interventions: Drug: Peginterferon alfa-2a

INTERVENTIONS:
Drug: Peginterferon alfa-2a — Patients will receive Peginterferon alfa-2a according to the standard medical practice

SUMMARY:
Patients will receive Peginterferon alfa-2a according to the standard medical practice but the observation period is 12 weeks

ELIGIBILITY:
Inclusion Criteria:

* History of HBsAg positive for more than 6 months
* HBeAg-positive or HBeAg-negative within 8 weeks
* Serum AST or ALT ≥ 80 IU/L
* HBe-Ag positive patients: Serum HBV DNA ≥ 1.0 X 10^5 copies/mL (or 20,000 IU/mL)
* HBeAg-negative patients: serum HBV DNA ≥ 1.0 X 10^4 copies/mL(or 2,000 IU/mL)

Exclusion Criteria:

* History of antiviral therapy for Chronic hepatitis B within 6 months of study enrollment
* Prior treatment of interferon
* Presence of viral coinfections (hepatitis C, hepatitis delta, or human immunodeficiency virus)
* Other chronic liver disease or decompensated liver disease
* platelet<90,000/mm3 or absolute neutrophil count < 1,500 mm3
* Pregnant or lactating woman
* History of Organ transplantation
* Treatment with immunosuppressive/immunomodulatory agents within 6 months prior to study entry

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 253 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-09 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
The proportion subjects with HBsAg ≤ 20,000 IU/mL at 12 week treatment of PEG-IFN in HBeAg-positive Chronic Hepatitis B | 12 week from baseline
The proportion subjects with any decline of HBsAg and/or HBV DNA decline more than 2 log copies/ml at 12 week treatment of PEG-IFN in HBeAg-negative CHB | 12 week from baseline

SECONDARY OUTCOMES:
The change of HBV DNA at Week 12 from baseline | 12 week from baseline
The change of HBsAg at Week 4, 8, 12 from baseline | 4, 8, 12 week from baseline
The change of ALT at week 4, 8, 12 from baseline | 4, 8, 12 week from baseline
The proportion of HBV DNA undetectable level (< 60 IU/mL, approximately 300 copies/mL) at week 12 | 12 week from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Sang Hoon Ahn, Principal Investigator — Severance Hospital
Locations (1):
- Severance Hospital, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No